CLINICAL TRIAL: NCT05542108
Title: Adding Motion to Contact: A New Model for Low-cost Family Centered Very-early Onset Intervention in Very Preterm-born Infants
Acronym: NTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Pisa (Other)
Collaborators: IRCCS Fondazione Stella Maris (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Andrea Guzzetta, Full Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NelleTueMani
Record Dates: First submitted 2022-09-08; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Premature Birth; Brain Injuries
Keywords: Early Intervention; Family-Centered Care; Neonatology; High-Risk Infant; Sensory Motor Stimulation; Maternal Voice; Tactile stimulation; Kinesthetic stimulation
MeSH Terms: conditions — Premature Birth; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Two intervention groups, Randomised Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes assessors are blind to the group assignment of the infant. Care provider (Parents and Research staff supporting parents in intervention can not be masked to the group assignment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensory Stimulation and Family Education Group (MSG) (Experimental): Parents of the MSG will be asked to carry out up to two treatment sessions per day with their child, until they reach the 8th post-term week. Sessions will initially be carried out together with a therapist who will have the task of transmitting the necessary skills to parents/caregivers.
  In addition, all families will receive the evidence-based program of Family Education which is based on the promotion of the parent-child relationship through the recognition of behavioral states, methods of interaction, facilitation strategies in the relationship.
  The family education group sessions involve about 6 meetings (1-2 a week) of 30-45 minutes that are carried out during the hospitalization in the NIC directly at the child's bed between the operator and one or both parents. Each meeting involves the discussion of one of the following topics.
  Interventions: Behavioral: Multisensory Stimulation and Family Education Group
- Family Education Only Group (FEG) (Active Comparator): Parents of the FEG group infants will be asked to participate in an evidence based program for parents of NICU infants that includes 6-8 visits with a a trained healthcare provider operator.
  This evidence-based program of early intervention based on the promotion of the parent-child relationship through the recognition of behavioral states, methods of interaction, facilitation strategies in the relationship.
  The program takes its conceptual basis from the Mother Infant Transaction Program (MITP).
  It involves about 6 meetings (1-2 a week) of 30-45 minutes that are carried out during the hospitalization in the NICU directly at the child's bed between the operator and one or both parents.
  Interventions: Behavioral: Family Education Only Group (FEG)

INTERVENTIONS:
Behavioral: Multisensory Stimulation and Family Education Group — Bedside intervention directly with infant with trained healthcare providers and parents. Includes two parts: twice daily multisensory stimulation sessions and separate family education meetings completed with individual infant parent/s and trained operator.
  Arms: Multisensory Stimulation and Family Education Group (MSG)
Behavioral: Family Education Only Group (FEG) — Bedside intervention directly with infant with trained healthcare providers and parents. Includes family education meetings completed with individual infant parent/s and trained operator.
  Arms: Family Education Only Group (FEG)

SUMMARY:
This project is a Randomised Clinical Trial that includes a tactile-kinesthetic somatosensory stimulation or family centred education intervention with families of preterm infants at risk for sensori-motor disorders.

This is a study will be based on the adaptation of the intervention previously described and published by Guzzetta and colleagues (2009), and will include an improved and increased kinesthetic component, to be performed in infants born very prematurely and preterm infants with a documented brain injury. The intervention will start in neonatology during the infant hospitalization and continue at the child's home until two months of correct age.

DETAILED DESCRIPTION:
Preterm babies, specifically with gestational age < 33+6 weeks, will be recruited and assigned (randomized) into an a Multisensory stimulation + Family Education Group (MSG) or a Family Education Only Group (FEG).

When the clinical condition of the child is stable and after a short training, parents of the MSG will be asked to carry out up to two treatment sessions per day with their child, until they reach the 8th post-term week. Sessions will initially be carried out together with a therapist who will have the task of transmitting the necessary skills to parents/caregivers. The therapist will assist parents through practical demonstrations, theoretical explanations and by answering the parents' questions.

The treatment will consist of sessions of approximately 25-30 minutes. The main purposes of the intervention will be clearly explained to the parents, and in particular the goal of maintaining a calm and natural interaction during the session.

In addition, all families will receive the evidence-based program of Family Education which is based on the promotion of the parent-child relationship through the recognition of behavioral states, methods of interaction, facilitation strategies in the relationship.

It takes its conceptual basis from the Mother Infant Transaction Program (MITP). It is a specific and re-adapted version for the preterm infant hospitalized in NICU

The family education group sessions involve about 6 meetings (1-2 a week) of 30-45 minutes that are carried out during the hospitalization in the NIC directly at the child's bed between the operator and one or both parents. Each meeting involves the discussion of one of the following topics.

ELIGIBILITY:
Inclusion Criteria:

* premature infants born <29 weeks of gestation age or premature infants (born < 33+6 weeks gestation age) with a documented brain injury .

Exclusion Criteria:

* Clinical instability, based on standard medical evaluation of preterm infants (eg: children with mechanical ventilation or under sedation)
* Genetic-malformative conditions

Ages: 1 Week to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
General Movements (GM) | 10-16 weeks corrected age
  The quality of general movements (based on standard observation of infant movements) will be assessed
Electroencephalogram (EEG) | 3 months corrected age
  The EEG inter-burst interval, asymmetries and global and local spectral power will be analysed

SECONDARY OUTCOMES:
Developmental outcome assessment | 12 months corrected age
  Bayley Scales of Infant Development Third Edition will be conducted including the Cognitive, Language (Receptive & Expressive), Motor (Gross & Fine), Social-Emotional and Adaptive sub scales. Each sub scale score will be calculated based on the age (months of age) of the infant at the time assessment. Higher scores mean a better outcome.

OTHER OUTCOMES:
Family well-being questionnaires | Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  The Infant Toddler Quality of Life QuestionnaireTM (ITQOL)
Family well-being questionnaire | Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  Edinburg Postnatal Depression Scale (EPDS)
Family well-being questionnaire | Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  Depression Anxiety Stress Scale (DASS-21)
Family well-being questionnaire | Before discharge from the Neonatal Unit (on average at 5 weeks post term age), 3, 6, 12 months corrected age
  Coping Orientation to Problems Experienced (COPE - NVI)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the Individual Participant Data